CLINICAL TRIAL: NCT05697848
Title: Pain Education: Treatment of Patients Affected by Chronic Low Back Pain, Randomized Controlled Study
Brief Title: Pain Education in Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Principal Investigator, Matteo Gallotta, Physiotherapist, Istituti Clinici Scientifici Maugeri SpA
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CE2556
Record Dates: First submitted 2023-01-13; First posted 2023-01-26 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Low Back Pain; Rehabilitation; Pain
MeSH Terms: conditions — Low Back Pain; Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Education group (Experimental): The patients of the experimental group will undergo pain education in addition to individual physiotherapy ( manual therapy and active exercises ).
  Interventions: Other: Physiotherapy combined with Pain Education
- Control group (Active Comparator): The patients of the control group will undergo individual physiotherapy ( manual therapy and active exercises ).
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy combined with Pain Education — Patients with chronic low back pain receive manual therapy treatment combined with Pain Education sessions.
  Arms: Pain Education group
Other: Physiotherapy — Patients with chronic low back pain receive manual therapy treatment
  Arms: Control group

SUMMARY:
The Pain Neuroscience Education (PNE) aims to reconceptualize pain from a marker of tissue damage to a marker of the perceived need to protect body tissue.

The purpose of this study is to verify the long-term efficacy (6 months) of a Pain Education treatment in patients with chronic low back pain, compared to a conventional treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Patients with low back pain of musculoskeletal origin for at least 3 months
* Patients free from NSAID and/or opioid analgesic therapy for at least 1 month
* Years of education: over 13
* Italian mother-tongue

Exclusion Criteria:

* Presence of neurological symptoms on provocative tests
* Recent surgical procedure
* Patients suffering from fibromyalgia or other rheumatological pathology
* Psychiatric pathologies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
NRS | Baseline
  Numeric Rating Scale. Score ranges from 0 (no pain) to 10 (the worst pain ever possible)
NRS | 4 weeks
  Numeric Rating Scale. Score ranges from 0 (no pain) to 10 (the worst pain ever possible)
NRS | 6 months
  Numeric Rating Scale. Score ranges from 0 (no pain) to 10 (the worst pain ever possible)
PCS | Baseline
  Pain Catastrophizing Scale. Score ranges from 0 to 52. Higher scores are associated with higher amounts of pain catastrophizing.
PCS | 4 weeks
  Pain Catastrophizing Scale. Score ranges from 0 to 52. Higher scores are associated with higher amounts of pain catastrophizing.
PCS | 6 months
  Pain Catastrophizing Scale. Score ranges from 0 to 52. Higher scores are associated with higher amounts of pain catastrophizing.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Scientifici Maugeri, Milan, Italy

IPD SHARING:
Plan to Share IPD: No